CLINICAL TRIAL: NCT05563493
Title: Comparison of the Effects of Chair-Based Exercise Training on Respiratory Functions, Exercise Capacity and Quality of Life in Patients With Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Brief Title: Effects of Chair-Based Exercise Training on Exercise Capacity in Patients With Acute Exacerbation of COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Zeynep Pelin Dündar, Research Assistant, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1
Record Dates: First submitted 2022-09-26; First posted 2022-10-03 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2022-09

CONDITIONS: Acute Exacerbation of COPD
Keywords: Chair-based exercise training
MeSH Terms: interventions — Control Groups; Breathing Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group, Chair-Based Exercise Training (Experimental): Treatment group will receive chair-based exercise training. Chair-based exercise training consisting of 20 different exercises will be applied in 2-3 sets with an average of 8-15 repetitions. Rest between sets will average 45-60 seconds.
  Interventions: Other: Treatment group, Chair-Based Exercise Training
- Control group, Breathing exercise (Other): Control group will receive breathing exercises.
  Interventions: Other: Control group, Breathing exercise

INTERVENTIONS:
Other: Treatment group, Chair-Based Exercise Training — The weights of the elastic bands to be used in the exercises will be determined by the physiotherapist according to the abilities and development of the participants.
  The intensity of the exercise will be adjusted according to the dyspnea or fatigue patients feel according to the Modified Borg Scale.
  During the exercises, heart rate and oxygen saturation will be measured with a pulse oximeter, and blood pressure will be measured with a sphygmomanometer.
  Chair-based exercise training will be applied to the patients every day they are hospitalized.
  Arms: Treatment group, Chair-Based Exercise Training
Other: Control group, Breathing exercise — Breathing exercise will be applied to the patients every day they are hospitalized.
  Arms: Control group, Breathing exercise

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is the leading cause of morbidity and mortality worldwide, a respiratory disease characterized by chronic airflow limitation that is not completely reversible.

Impaired pulmonary functions, decreased exercise capacity and quality of life and increased dyspnea perception is prevalent in patients with acute exacerbations of COPD.It was demonstrated exercise training has beneficial effects in patients with acute exacerbations of COPD.

The purpose of this study to evaluate the effects of chair-based exercise training on exercise capacity, respiratory functions, dyspnea, balance, depression anxiety and quality of life in COPD patients in acute exacerbation.

DETAILED DESCRIPTION:
Acute exacerbations of COPD are generally defined as events in the natural course of the disease characterized by a change in the patient's initial dyspnea, cough or sputum beyond normal daily variations. The main consequences of COPD in acute exacerbation are increased mortality, deterioration in health-related quality of life, faster decline in lung function, marked reduction in physical activity and worsening of peripheral muscle weakness, which have a direct impact on patients' health. Although exacerbations are diagnosed based on respiratory symptoms, there is evidence that they have systemic consequences, including a detrimental effect on skeletal muscle function, exercise tolerance and quality of life.

Chair-based exercise training is defined as a structured and progressive exercise program applied by trainers that provides stability using a chair, which is a part of exercise training for the elderly. It is thought that it would be beneficial to study such an exercise program, since COPD patients in acute exacerbation have less mobilization during hospitalization.

In a limited number of studies, some inconsistencies were observed in the exercises of patients with acute exacerbation of COPD. Studies can therefore now focus on investigating comparisons between different intervention lengths, session durations and frequencies, and intensities of exercise training. For this reason, in our planned study, we will investigate the effects of chair-based exercise training in COPD patients in acute exacerbation. There is no study in the literature investigating the effects of chair-based exercise training in COPD patients in acute exacerbation. For this reason, our study will provide important information support to the literature.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were hospitalized due to acute exacerbation of COPD

Exclusion Criteria:

* Patients with orthopedic or neurological problems that may interfere with assessment and education,
* Uncooperative patients,
* Patients with advanced heart problems such as acute coronary syndrome, stable angina pectoris, severe arrhythmias (Atrial fibrillation etc.), decompensated heart failure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-08-20 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Functional Exercise Capacity | Seven day
  Functional exercise capacity will be evaluated with 6-minute walk test.
Pulmonary Function Test | Seven day
  This test was evaluated using a spirometry by which is evaluated dynamic lung functions expressed as percentages of expected values.

SECONDARY OUTCOMES:
Dyspnea | Seven day
  The severity of dyspnea during daily living activities is evaluated using the Modified Medical Research Council (MMRC) dyspnea scale.
One Minute Sit to Stand Test | Seven day
  The number of completed sit to stand repetitions in 1 minute. Patients stand/sit from a chair as many times as they can in one minute.
Timed Up and Go Test | Seven day
  The Timed Up and Go test is evaluated dynamic balance.
Depression and Anxiety | Seven day
  Evaluated using Hospital Anxiety and Depression Scale (Turkish versions of all scales)
Life of quality | Seven day
  Saint George's Respiratory Questionnaire (SGRQ) (Turkish versions of all scales) is used to assess the quality of life of COPD patients.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Pelin DÜNDAR, MSc,PT, Principal Investigator — Necmettin Erbakan University; Nihan KAFA, Study Director — Gazi University; Hülya VATANSEV, Study Director — Necmettin Erbakan University; Neslihan DURUTÜRK, Study Chair — Baskent University; Adil ZAMANİ, Study Chair — Necmettin Erbakan University
Locations (1):
- Necmettin Erbakan University Nezahat Keleşoğlu Faculty of Health Sciences, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liao S, Wang F, Lin Q, Jian F, Li Y, Zhong Q, Huang Y, Lin Y, Wang H. Effect of sitting and lying Liuzijue exercise for pulmonary rehabilitation in acute exacerbation of chronic obstructive pulmonary disease patients with non-invasive ventilation: a randomized controlled trial. Ann Palliat Med. 2021 Sep;10(9):9914-9926. doi: 10.21037/apm-21-2157. PMID 34628916
- [Background] Knaut C, Bonfanti Mesquita C, Dourado VZ, de Godoy I, Tanni SE. Evaluation of Inflammatory Markers in Patients Undergoing a Short-Term Aerobic Exercise Program while Hospitalized due to Acute Exacerbation of COPD. Int J Inflam. 2020 Apr 28;2020:6492720. doi: 10.1155/2020/6492720. eCollection 2020. PMID 32411343
- [Background] Burtin C, Decramer M, Gosselink R, Janssens W, Troosters T. Rehabilitation and acute exacerbations. Eur Respir J. 2011 Sep;38(3):702-12. doi: 10.1183/09031936.00079111. Epub 2011 Jun 30. PMID 21719481
- [Background] Kon SS, Canavan JL, Man WD. Pulmonary rehabilitation and acute exacerbations of COPD. Expert Rev Respir Med. 2012 Nov;6(5):523-31; quiz 531. doi: 10.1586/ers.12.47. PMID 23134247